CLINICAL TRIAL: NCT07311577
Title: Disitamab Vedotin Combined With Platinum and Bevacizumab as First-Line and Maintenance Therapy for HER2-Expressing, HRD-Negative High-Risk Ovarian Cancer: A Multicenter, Non-Randomized, Single-Arm Phase II Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Xiaoxiang Chen, Professor, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDTYPEC170
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer Metastatic; Ovarian Cancer Metastatic Recurrent
Keywords: RC48; HRD-Negative High-Risk Ovarian Cancer; HER2-expressing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: RC48+Carboplatin+Bevacizumab

INTERVENTIONS:
Drug: RC48+Carboplatin+Bevacizumab — First-line phase:Carboplatin AUC 5 intravenously on Day 1 every 21 days over 1 h; Bevacizumab 7.5-15 mg/kg intravenously on Day 1 every 21 days over 30-90 min. Maintenance phase:Patients who achieve response (CR or PR) will continue disitamab vedotin monotherapy plus bevacizumab (investigator decides whether to continue disitamab vedotin and for how long).
  Maintenance duration: bevacizumab until disease progression or up to 22 cycles; disitamab vedotin up to 6 months (8 cycles).

SUMMARY:
This is a prospective, multicenter, phase II study designed to evaluate the efficacy and safety of disitamab vedotin combined with platinum plus bevacizumab as first-line therapy for HER2-expressing, HRD-negative high-risk ovarian cancer. Forty-three patients with pathologically confirmed HRD-negative high-risk ovarian cancer will be enrolled. After enrollment, patients will receive disitamab vedotin plus platinum and bevacizumab as first-line and maintenance treatment.

First-line phase:

Carboplatin AUC 5 intravenously on Day 1 every 21 days over 1 h ,Bevacizumab 7.5-15 mg/kg intravenously on Day 1 every 21 days over 30-90 min.

Maintenance phase:

Patients who achieve response (CR or PR) will continue disitamab vedotin monotherapy plus bevacizumab (investigator decides whether to continue disitamab vedotin and for how long).

Maintenance duration: bevacizumab until disease progression or up to 22 cycles; disitamab vedotin up to 6 months (8 cycles).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation with written informed consent.
* Age 18-75 years.
* Expected survival ≥ 12 weeks.
* Histologically/cytologically confirmed advanced ovarian carcinoma (FIGO Stage III-IV).
* HRD-negative status per local assessment.
* High-risk features: macroscopic residual disease after primary cytoreductive surgery for Stage III; prior neoadjuvant chemotherapy; or Stage IV disease.
* ≥ 1 RECIST v1.1 measurable lesion (long-axis ≥ 10 mm by spiral CT or ≥ 15 mm short-axis for lymph nodes).
* HER2 expression documented locally (IHC 1+, 2+, or 3+); archival or fresh tumor tissue (paraffin block or unstained slides) must be available for central confirmation.
* ECOG performance status 0-1.
* Adequate organ function within 14 days before enrolment (no transfusion/haematinics/G-CSF allowed):

Haematology

1. Hb ≥ 90 g/L
2. WBC ≥ 3 × 10⁹/L
3. ANC ≥ 1.5 × 10⁹/L
4. PLT ≥ 90 × 10⁹/L Biochemistry

a) TBIL ≤ 1.5 × ULN b) ALT/AST/ALP ≤ 3 × ULN (≤ 5 × ULN if liver metastases) c) Serum creatinine ≤ 1.5 × ULN or CrCl ≥ 60 mL/min (Cockcroft-Gault)

* Urinalysis: dipstick proteinuria < 2+ or 24-h urine protein < 1 g.
* Cardiac function: NYHA class < III and LVEF ≥ 50 % by echocardiography. -
* Women must be surgically sterile, post-menopausal, or use an approved contraceptive method from screening until 6 months after the last dose; serum pregnancy test negative within 7 days of first dose and not breastfeeding.
* Able and willing to comply with all study and follow-up procedures.

Exclusion Criteria:

* Non-high-risk histologic sub-types of ovarian carcinoma.
* CNS metastases and/or carcinomatous meningitis. -
* Requirement for parenteral hydration/nutrition OR clinical/radiologic evidence of partial bowel obstruction or perforation.
* ≥ Grade-2 peripheral neuropathy. -
* Active bleeding or high bleeding-risk conditions (e.g., known coagulopathy, tumour encasing major vessels).
* Interval between cytoreductive surgery and first bevacizumab dose < 28 days.
* Concurrent malignancy or history of another primary malignancy within 5 years (except adequately treated in-situ cervix cancer, basal- or squamous-cell skin cancer).
* Major surgery within 4 weeks before first study dose and not fully recovered.
* Symptomatic or medically-requiring large-volume pleural effusion or ascites. - Live-attenuated vaccine within 30 days before first dose or planned during study.
* Significant arterial/venous thrombo-embolic or cerebro-cardiovascular event within 12 months before screening (e.g., DVT, PE, cerebral infarction, intracranial haemorrhage, MI); asymptomatic calf-muscle DVT not needing intervention or lacunar infarct without sequelae are allowed.
* Uncontrolled systemic diseases judged by investigator: diabetes, liver cirrhosis Child-Pugh B/C, interstitial pneumonitis, severe COPD, etc.
* Clinically-relevant cardiovascular disorders:

  1. PR interval > 0.24 s or 2nd/3rd-degree AV block.
  2. Uncontrolled hypertension (SBP > 150 mmHg or DBP > 90 mmHg).
  3. MI, unstable angina or significant arrhythmia < 6 months before enrolment.
  4. NYHA class ≥ II congestive heart failure.
  5. Serious arrhythmia requiring anti-arrhythmic therapy.
  6. ≥ Stage-II peripheral vascular disease (except transient ischaemia < 24 h without permanent deficit and no surgery).
  7. Cerebrovascular accident within 6 months.
* Severe infection within 4 weeks before first dose (IV antibiotics/antifungals/ antivirals required) or unexplained fever > 38.5 °C during screening; major surgery within 3 weeks.
* Active autoimmune or immunodeficiency disorders (e.g., autoimmune hepatitis, interstitial pneumonia, uveitis, RA, IBD, hypophysitis, vasculitis, nephritis). Exceptions: stable hypothyroidism on replacement, type-1 diabetes well controlled with insulin.
* Autoimmune disease requiring systemic immunosuppressive/immunomodulatory therapy within 2 years before first dose (stable replacement therapy with thyroxine, insulin or physiological corticosteroids permitted).
* Active or poorly controlled infection, including:

  1. HIV positive (HIV-1/2 antibody).
  2. Active hepatitis B (HBsAg positive or HBV DNA > 2 000 IU/mL with abnormal LFT).
  3. Active hepatitis C (HCV antibody positive or HCV RNA ≥ 10³ copies/mL with abnormal LFT).
  4. Active tuberculosis.
  5. Other uncontrolled infection > CTCAE v5.0 grade 2.
* History of other malignancy within 5 years (except adequately treated in-situ cervical cancer or basal/squamous-cell skin cancer). -
* Concurrent participation in another interventional clinical trial or investigational agent/device within 4 weeks before first dose. -
* Known hypersensitivity or intolerance to study drugs or their excipients. -
* History of substance abuse that cannot be abstained from, or any psychiatric disorder that may interfere with compliance.

Any other condition that, in the investigator's opinion, could increase risk or preclude safe completion of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment until 16 months
  From enrollment until documented disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 weeks
  Disease Control Rate (DCR) is defined as the proportion of patients who achieve a Best Overall Response of PR or CR .
Disease Control Rate (DCR) | up to 24 weeks
  Disease Control Rate (DCR) is defined as the proportion of patients who achieve a Best Overall Response of PR or CR or SD.
overall survival（OS） | Up to 5 years
  From enrollment until death from any cause.
Incidents of Adverse Events | 30 days after the end of treatment
  All patients who receive at least one dose of any study drug are included in the safety-analysis set.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided